CLINICAL TRIAL: NCT05903807
Title: [68Ga]Ga-FAPI-46 PET/CT: the Diagnostic Accuracy for Primary Staging and Re-staging of Patients with Ovarian Cancer
Brief Title: [68Ga]Ga-FAPI-46 PET/CT in Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Morten Bentestuen, Principal Investigator, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EU CT nr: 2023-505938-98-00
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: Cancer; FAPI; FAPI PET/CT; Fibroblast activation protein inhibitor; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — FAPI-46

STUDY DESIGN:
Intervention Model Description: Fifty consecutive patients newly diagnosed with ovarian cancer are recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ovarian cancer or high risk of ovarian cancer (Experimental): Patients with newly diagnosed ovarian cancer or high risk of ovarian cancer undergo FAPI PET/CT in addition to conventional imaging
  Interventions: Drug: 68Ga-FAPi-46

INTERVENTIONS:
Drug: 68Ga-FAPi-46 — Ovarian cancer patients undergo 68Ga-FAPI-46 at primary staging and at restaging

SUMMARY:
Fifty (n=50) patients with newly diagnosed ovarian cancer will undergo FAPI PET/CTs in addition to routine diagnostic workup (including FDG PET/CT) at primary staging and restaging.

The FAPI PET/CT results will be compared to conventional imaging (including FDG PET/CT) using histopathology as reference standard, and the diagnostic accuracy will be determined. FAP-immunohistochemistry will be conducted in surgical specimens. FAPI PET/CT's impact on patient management and the prognostic value of FAPI PET/CT will be evaluated.

DETAILED DESCRIPTION:
A new and promising PET-tracer in oncology has been developed; Gallium-68 labelled fibroblast activation protein inhibitor (FAPI). In general, FAPI PET/CT delivers increased sensitivity compared to 18F-Fluorodeoxyglucose (FDG) PET/CT in cancer types of mesenchymal origin (i.e., sarcomas), and in cancers characterized by a large proportion of stromal cells such as gastric and pancreatic cancers. It is currently debated whether FAPI PET/CT will take over FDG PET/CTs well-established role in oncological PET/CT, but more studies are needed to evaluate the diagnostic accuracy. The clinical interest in FAPI extends beyond the use as a diagnostic tool, as the 68Ga-isotope can be replaced by a β-emitting isotope, e.g., 177-Lu or 90-Y, enabling radionuclide therapy of FAPI-avid cancers.

Not long after the development of FAPI, the clinical value of FAPI PET/CT in ovarian cancer patients was highlighted by several case reports where FAPI PET/CT detected far more peritoneal metastases than FDG PET/CT. Only recently have cohort studies in ovarian cancer been conducted. In these studies, FAPI PET/CT demonstrates promising results when compared to FDG PET/CT, especially in peritoneal lesions.

Even though the results of FAPI PET/CT compared to conventional imaging seem convincing, there are several limitations and therefore FAPI PET/CT is not yet implemented in cancer diagnostics.

The investigators are conducting a prospective explorative study complying with the Standard for Reporting Diagnostic Accuracy (STARD) criteria where 50 patients with ovarian cancer are recruited.

Study subject will undergo FAPI PET/CT at primary staging (before treatment, i.e., neoadjuvant chemotherapy or surgery) and at restaging (after neoadjuvant chemotherapy - before surgery) in addition to routing diagnostic workup (including FDG PET/CT). The FAPI PET/CT will be blinded and the choice of treatment will not be influence by the FAPI PET/CT results'. The additional scans will not interfere with or delay routine diagnostic workup or treatment. The FAPI PET/CTs (at primary staging and restaging) will be compared to the corresponding FDG PET/CTs, and histopathology of biopsied material and surgical specimens will serve as reference standard. FAPI PET/CTs before and after neoadjuvant chemotherapy will be assessed and compared to the FDG PET/CTs. FAP-immunohistochemistry will be conducted in surgical specimens. A tentative retrospective Multi-Disciplinary Team conference (MDT) will be arranged where treating clinicans are presented the FAPI PET/CT, and potential changes in patient management will be evaluated. This tentative MDT will not influence patient management. Follow up will be conducted for 10 years to evaluate the prognostic value of FAPI PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with biopsy verified ovarian cancer or highly suspected to have ovarian cancer (based on all data presented at the gynecological cancer MDT) and referred to primary staging with FDG PET/CT
* Deemed resectable and operable at the MDT with or without neoadjuvant chemotherapy
* Considered physically and mentally able to participate in the research project
* 18-years or older and able to consent to project participation
* Can read and understand Danish

Exclusion Criteria:

* Patients with non-resectable, inoperable, or recurrent ovarian cancer
* Patients with an imminent need for surgery or in an emergency
* Known concurrent other malignancy within the previous 5 years other than non-melanoma skin cancer
* Patients not suited for surgery or neoadjuvant chemotherapy followed by surgery
* Subject weighing more than 180 kg (weight limit scanner) or unable to fit within the imaging gantry
* History of allergic reactions / hypersensitivity attributed to 18F-FDG or 68Ga-FAPI-46.
* Severe claustrophobia unresponsive to oral anxiolytics
* Subjects with any medical condition or other circumstances that, in the opinion of the Investigator, would significantly decrease the reliability of data, achievement of study objectives or completing the study.
* Pregnant, lactating, or breastfeeding women.
* Potential pregnant women of childbearing potential [1] not using effective contraceptives [2]. Potential pregnancy will be ascertained by a pregnancy test (urine humane choriogonadotropin (HCG)) or serum b-HCG within 48 hours prior to the FAPI PET/CT.
* Inability to remain still for the duration of the examination

  1. Women of childbearing potential are defined as all women physiologically capable of becoming pregnant, i.e., not sterilized (bilateral tubectomy/occlusion, hysterectomy, bilateral oophorectomy) and not post-menopausal. In cases of uncertain menopausal status, serum follicle stimulating hormone (FSH) levels and menstruation history can be assessed
  2. Effective contraceptives include sexual abstinence, vasectomized partner, combined hormonal contraception (oral, intravaginal, transdermal), progesterone-only contraceptive (oral, injectable, implantable), or working intrauterine device (hormonal, non-hormonal).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 2 years
  Diagnostic accuracy Compare the FAPI PET/CT and FDG PET/CT findings in primary tumor, regional lymph nodes and distant metastases to a histopathological reference standard where the sensitivity, specificity, positive predicative value, and negative predicative values of the PET/CTs are determined, both at primary staging and at restaging
Staging | 2 years
  Compare the cancer stage as determined by FAPI PET/CT compared to conventional imaging (including FDG PET/CT) at primary staging and at restaging (after neoadjuvant chemotherapy). The proportion of patients downstaged, unchanged stage, and upstaged, due to the added FAPI PET/ CT are determined.
Patient management | 2 - 2.5 years
  Investigate what proportion of patients will be (hypothetically) treated differently due to an added FAPI PET/CT at primary staging and at restaging (after neoadjuvant chemotherapy) by the treating clinicians

SECONDARY OUTCOMES:
Uptake values | 2 years
  Standardized uptake value (SUV) and tumor-to-background ratio (TBR) values for primary, regional lymph nodes, and distant metastases for FAPI PET/CT and compare these values to FDG PET/CT, both at primary staging and at restaging (after neoadjuvant chemotherapy)
Chemotherapy effect on uptake values | 2 - 2.5 years
  Changes in SUV and TBR in primary, regional lymph nodes, and distant metastases for FAPI PET/CT - from before to after neoadjuvant chemotherapy and compare these values to the FDG PET/CT parameters.
Unexpected 68Ga-FAPI-46 PET/CT findings | 1-2 years
  Seek supplementary information in medical records, biochemistry, pathology, or other imaging modalities for a final diagnosis/condition in cases of unexpected FAPI PET/CT findings not related to the known cancer
Interobserver readability | 4 years
  Conduct an interobserver study of FAPI PET/CTs performed in the present and other future FAPI PET/CT in cancers studies.
Prognostic value | 10 years
  Investigate the prognostic value of FAPI PET/CT versus FDG PET/CT by conducting a 10 years follow up on included cancer patients. Overall survival (OS) and Recurrence free survival (RFS) will be estimated

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Lindner T, Loktev A, Altmann A, Giesel F, Kratochwil C, Debus J, Jager D, Mier W, Haberkorn U. Development of Quinoline-Based Theranostic Ligands for the Targeting of Fibroblast Activation Protein. J Nucl Med. 2018 Sep;59(9):1415-1422. doi: 10.2967/jnumed.118.210443. Epub 2018 Apr 6. PMID 29626119
- [Background] Kessler L, Ferdinandus J, Hirmas N, Bauer S, Dirksen U, Zarrad F, Nader M, Chodyla M, Milosevic A, Umutlu L, Schuler M, Podleska LE, Schildhaus HU, Fendler WP, Hamacher R. 68Ga-FAPI as a Diagnostic Tool in Sarcoma: Data from the 68Ga-FAPI PET Prospective Observational Trial. J Nucl Med. 2022 Jan;63(1):89-95. doi: 10.2967/jnumed.121.262096. Epub 2021 Apr 30. PMID 33931468
- [Background] Rohrich M, Naumann P, Giesel FL, Choyke PL, Staudinger F, Wefers A, Liew DP, Kratochwil C, Rathke H, Liermann J, Herfarth K, Jager D, Debus J, Haberkorn U, Lang M, Koerber SA. Impact of 68Ga-FAPI PET/CT Imaging on the Therapeutic Management of Primary and Recurrent Pancreatic Ductal Adenocarcinomas. J Nucl Med. 2021 Jun 1;62(6):779-786. doi: 10.2967/jnumed.120.253062. Epub 2020 Oct 23. PMID 33097632
- [Background] Dendl K, Schlittenhardt J, Staudinger F, Kratochwil C, Altmann A, Haberkorn U, Giesel FL. The Role of Fibroblast Activation Protein Ligands in Oncologic PET Imaging. PET Clin. 2021 Jul;16(3):341-351. doi: 10.1016/j.cpet.2021.03.012. PMID 34053578
- [Background] Qin C, Song Y, Gai Y, Ruan W, Liu Q, Liu F, Zheng D, Zhang P, Liu H, Zhang T, Tao K, Lan X. Gallium-68-labeled fibroblast activation protein inhibitor PET in gastrointestinal cancer: insights into diagnosis and management. Eur J Nucl Med Mol Imaging. 2022 Oct;49(12):4228-4240. doi: 10.1007/s00259-022-05847-0. Epub 2022 Jun 3. PMID 35657428
- [Background] Meyer C, Dahlbom M, Lindner T, Vauclin S, Mona C, Slavik R, Czernin J, Haberkorn U, Calais J. Radiation Dosimetry and Biodistribution of 68Ga-FAPI-46 PET Imaging in Cancer Patients. J Nucl Med. 2020 Aug;61(8):1171-1177. doi: 10.2967/jnumed.119.236786. Epub 2019 Dec 13. PMID 31836685
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Zheng W, Liu L, Feng Y, Wang L, Chen Y. Comparison of 68 Ga-FAPI-04 and fluorine-18-fluorodeoxyglucose PET/computed tomography in the detection of ovarian malignancies. Nucl Med Commun. 2023 Mar 1;44(3):194-203. doi: 10.1097/MNM.0000000000001653. Epub 2022 Dec 7. PMID 36472415
- [Background] Liu S, Feng Z, Xu X, Ge H, Ju X, Wu X, Song S. Head-to-head comparison of [18F]-FDG and [68 Ga]-DOTA-FAPI-04 PET/CT for radiological evaluation of platinum-sensitive recurrent ovarian cancer. Eur J Nucl Med Mol Imaging. 2023 Apr;50(5):1521-1531. doi: 10.1007/s00259-022-06096-x. Epub 2023 Jan 10. PMID 36624168
- [Background] Dendl K, Koerber SA, Finck R, Mokoala KMG, Staudinger F, Schillings L, Heger U, Rohrich M, Kratochwil C, Sathekge M, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI-PET/CT in patients with various gynecological malignancies. Eur J Nucl Med Mol Imaging. 2021 Nov;48(12):4089-4100. doi: 10.1007/s00259-021-05378-0. Epub 2021 May 29. PMID 34050777
- [Background] Xi Y, Sun L, Che X, Huang X, Liu H, Wang Q, Meng H, Miao Y, Qu Q, Hai W, Li B, Feng W. A comparative study of [68Ga]Ga-FAPI-04 PET/MR and [18F]FDG PET/CT in the diagnostic accuracy and resectability prediction of ovarian cancer. Eur J Nucl Med Mol Imaging. 2023 Jul;50(9):2885-2898. doi: 10.1007/s00259-023-06235-y. Epub 2023 Apr 24. PMID 37093313
- [Derived] Bentestuen M, Ladekarl M, Knudsen A, Zacho HD. Diagnostic accuracy and clinical value of [68Ga]Ga-FAPI-46 PET/CT for staging patients with ovarian cancer: study protocol for a prospective clinical trial. BMC Cancer. 2024 Jun 7;24(1):699. doi: 10.1186/s12885-024-12461-w. PMID 38849741